CLINICAL TRIAL: NCT05537896
Title: Prospective Evaluation of Xerava™ (Eravacycline) Prophylaxis in Hematological Malignancy Patients With Prolonged Neutropenia
Brief Title: Prospective Evaluation of Xerava Prophylaxis in Hematological Malignancy Patients With Prolonged Neutropenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Aaron Cumpston, PharmD, BCOP, Pharmacy Clinical Specialist, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2206591296
Record Dates: First submitted 2022-09-12; First posted 2022-09-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hematological Malignancy; Neutropenia
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia | interventions — eravacycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eravacycline (Experimental): Eravacycline- 1 mg/kg actual body weight IV Infusion over 60 minutes every 12 hours. Alternative dosing strategy 1.5mg/kg every 12 hourse.
  Interventions: Drug: Eravacycline

INTERVENTIONS:
Drug: Eravacycline — Eravacycline will be continued until one of the following criteria is met:
  * neutrophil recovery (ANC >500, post-nadir)
  * febrile neutropenia
  * breakthrough infection
  * any grade 3-4 toxicity related to eravacycline use
  * 21 days of therapy (maximum duration allowed per study protocol)
  Other Names: Xerava

SUMMARY:
Antibacterial prophylaxis is recommended in patients at high risk of infection, specifically patients undergoing acute leukemia induction therapy or hematopoietic stem cell transplant (HSCT) who are expected to have profound neutropenia (ANC<100 neutrophils/milliliter) for more than seven days. Xerava™ (eravacycline) has a broad spectrum of activity including many multi-drug resistant strains of bacteria. It is not an agent used for treatment of febrile neutropenia, making eravacycline a very attractive alternative to consider in this prophylactic setting. Eravacycline has activity against MRSA, VRE, and Clostridioides difﬁcile, all of which are common problems in this patient population. It also covers the majority of enteric gram-negative pathogens while also producing satisfactory tissue penetration and adequate plasma concentrations, which has classically been a concern with prior agents. Eravacycline has activity against coagulase-negative staphylococcus, which is a common catheter-related infection in leukemia and HSCT patients. The primary objective will be report the incidence of breakthrough infections during eravacycline prophylaxis for hematologic malignancy patients with prolonged neutropenia.

DETAILED DESCRIPTION:
Antibacterial prophylaxis is recommended in patients at high risk of infection, specifically patients undergoing acute leukemia induction therapy or hematopoietic stem cell transplant (HSCT) who are expected to have profound neutropenia (ANC<100 neutrophils/milliliter) for more than seven days.

Xerava™ (eravacycline) is a synthetic halogenated tetracycline class antibiotic, with a broad spectrum of activity including many multi-drug resistant strains of bacteria. It is not an agent used for treatment of febrile neutropenia, making eravacycline a very attractive alternative to consider in this prophylactic setting. Adverse effects with this agent are minimal including infusion site reactions and gastrointestinal disorders. Eravacycline has activity against MRSA, VRE, and Clostridioides difﬁcile, all of which are common problems in this patient population. It also covers the majority of enteric gram-negative pathogens while also producing satisfactory tissue penetration and adequate plasma concentrations, which has classically been a concern with prior agents. Eravacycline has activity against coagulase-negative staphylococcus, which is a common catheter-related infection in leukemia and HSCT patients. The primary objective will be report the incidence of breakthrough infections during eravacycline prophylaxis for hematologic malignancy patients with prolonged neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving induction chemotherapy for treatment of acute leukemia or receiving preparative regimen for HSCT
* Patient must provide informed consent.
* Bilirubin ≤ 3 x the ULN and AST/ALT ≤ 5 x ULN

Exclusion Criteria:

* Uncontrolled bacterial, viral or fungal infection at the time of study enrollment.
* Urinary tract infection receiving active treatment
* Acute pancreatitis (not necessary to work-up unless symptomatic)
* History of known hypersensitivity to eravacycline, tetracycline, doxycycline, minocycline, tigecycline, sarecycline, oxytetracycline, or omadacycline
* Pseudomonas infection within 30 days prior to study enrollment
* Receiving strong inhibitors or inducers of cytochrome P450 3A4 will be excluded from the study (see Appendix B for complete list of medications)
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Documented Breakthrough Infections | Up to 21 days
  Number of Incidences documented that subjects had a confirmed breakthrough infection.

SECONDARY OUTCOMES:
Adverse Events | Daily during Eravacycline
  Incidence of Adverse Events: CTCAE criteria. CTCAE stands for Common Terminology Criteria for Adverse Events; these criteria are also called "common toxicity criteria." In CTCAE, an adverse event (AE) is defined as any abnormal clinical finding temporally associated with the use of a therapy for cancer; causality is not required. These criteria are used for the management of chemotherapy administration and dosing, and in clinical trials to provide standardization and consistency in the definition of treatment-related toxicity.
Infection-related mortality | Up to 30 days
  Incidence of Infection-related mortality. Infection-related mortality is defined as any death that occurred in the presence of clinical or microbiological documented infection
All-cause mortality | Up to 30 days
  Incidence of All-cause mortality defined as any death occurring during the clinical trial period.
Acute GVHD | Up to 100 days
  Incidence of Acute Graft vs Host Disease (GVHD). GVHD is a complication of a bone marrow or stem cell transplant in which cells from a donor attack the tissues of the recipient.
Neutropenic fever | Up to 21 days
  Rate of neutropenic fever: Defined as development of febrile neutropenia (temperature >38.2 degrees C and ANC is <500 cells/mm3).
Time to neutropenic fever | Up to 21 days
  Time to development of febrile neutropenia (temperature >38.2 degrees C and ANC is <500 cells/mm3).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cumpston, PharmD, BCOP, Principal Investigator — West Virginia University
Locations (1):
- Aaron Cumpston, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No